CLINICAL TRIAL: NCT06909058
Title: Postoperative Restrictions for Patients Undergoing Minimally Invasive Gynecologic Procedures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Frappaolo (Other)
Responsible Party: Sponsor-Investigator, Anna Frappaolo, OBGYN Resident Physician, Women and Infants Hospital of Rhode Island
Organization: Women and Infants Hospital of Rhode Island (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2221729
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Care; MIGS
Keywords: postoperative care; minimally invasive gynecologic surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control. Patients to receive standard postoperative instructions. (No Intervention): Participants in the control group will receive standard postoperative instructions which would be given whether the patient was enrolled in this study or not. This includes written and verbal instructions not to lift anything heavier than 10 pounds, or partake in rigorous exercise (weightlifting, sit-ups) for at least 2 weeks postoperatively.
- Study. Patients to receive liberalized postoperative instructions. (Experimental): Participants in the study group will receive liberal postoperative instructions. This includes written and verbal instructions to resume normal activities of daily living without restriction at the discretion of the patient.
  Interventions: Behavioral: Study Postoperative Care

INTERVENTIONS:
Behavioral: Study Postoperative Care — The study group will be given general postoperative instructions. They will also receive liberal activity restrictions instructing the patient to resume normal activities of daily living at their own discretion without specific restrictions.
  Arms: Study. Patients to receive liberalized postoperative instructions.

SUMMARY:
The goal of this randomized controlled trial is to assess recovery in patients undergoing benign laparoscopic gynecologic surgery. The main question it aims to answer is: do liberalized postoperative restrictions improve patient recovery after laparoscopic gynecologic surgery?

Researchers will compare postoperative recovery surveys from the control group (patients given standard postoperative restrictions limiting activity for 2 weeks) to the research group (patients given liberalized postoperative instructions allowing them to engage in their normal activities of daily life at their own discretion without prescribed activity restrictions) to see if liberalized postoperative restrictions improve the recovery experience.

Participants will be asked to fill out a brief questionnaire at two time intervals, 1 week after surgery and 2 weeks after surgery.

DETAILED DESCRIPTION:
The questionnaire will consist of the Recovery Index-10 (RI-10), a short recovery-specific instrument to assess subjective postoperative recovery that is specifically validated for gynecologic surgery. It is graded on a 5-point numerical Likert scale ranging from "full disagreement" to "full agreement." The questionnaire asks questions regarding pain, stamina/ability to complete daily chores, energy, and sleep.

In addition to the RI-10 survey, a few additional questions will be asked to assess whether the patient has dependents they are responsible for, if they have returned to work, and if they have resumed driving.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* English speaking (Spanish speaking to be added once appropriate forms are professionally translated and approved)
* 5-8 mm port sites used during the surgery

Exclusion Criteria:

* Less than 18 years of age
* Primary language other than English (or Spanish once forms are professionally translated and approved)
* Use of port size >8mm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative recovery | The RI-10 will be completed by the patient at two time points: 1 week post-surgery, and 2 weeks post-surgery
  Postoperative recovery will be evaluated using the Recovery Index-10 (RI-10), a recovery-specific instrument to assess subjective postoperative recovery that is specifically validated for gynecologic surgery. It is graded on a 5-point numerical Likert scale ranging from "full disagreement" to "full agreement." The questionnaire asks questions regarding pain, stamina/ability to complete daily chores, energy, and sleep. Prior literature on the use and validation of RI-10 suggests a standard deviation of 20 and an effect size of 15.

SECONDARY OUTCOMES:
Postoperative complications | Within 2 weeks postoperatively
  Postoperative complications as defined by unscheduled patient contacts for pain or incisional complaints. This could include: ER visits, urgent clinic visits, phone calls regarding incisional complaints, any 30-day readmissions.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Foley, MD, Principal Investigator — Care New England - Women and Infants Hospital
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brolmann HA, Vonk Noordegraaf A, Bruinvels DJ, de Vet RH, Dirksz AA, Huirne JA. Can prolonged sick leave after gynecologic surgery be predicted? An observational study in The Netherlands. Surg Endosc. 2009 Oct;23(10):2237-41. doi: 10.1007/s00464-008-0287-0. Epub 2009 Jan 1. PMID 19118421
- [Result] Kluivers KB, Hendriks JC, Mol BW, Bongers MY, Vierhout ME, Brolmann HA, de Vet HC. Clinimetric properties of 3 instruments measuring postoperative recovery in a gynecologic surgical population. Surgery. 2008 Jul;144(1):12-21. doi: 10.1016/j.surg.2008.03.027. Epub 2008 May 21. PMID 18571580
- [Result] Min J, Kim JY, Ryu J, Park S, Courneya KS, Ligibel J, Kim SI, Jeon JY. Early Implementation of Exercise to Facilitate Recovery After Breast Cancer Surgery: A Randomized Clinical Trial. JAMA Surg. 2024 Aug 1;159(8):872-880. doi: 10.1001/jamasurg.2024.1633. PMID 38837150
- [Result] Mueller MG, Lewicky-Gaupp C, Collins SA, Abernethy MG, Alverdy A, Kenton K. Activity Restriction Recommendations and Outcomes After Reconstructive Pelvic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2017 Apr;129(4):608-614. doi: 10.1097/AOG.0000000000001924. PMID 28277355
- [Result] Arunachalam D, Heit MH. Impact of postoperative instructions on physical activity following pelvic reconstructive surgery: a randomized controlled trial. Int Urogynecol J. 2020 Jul;31(7):1337-1345. doi: 10.1007/s00192-020-04239-y. Epub 2020 Feb 15. PMID 32062677
- [Result] Weir LF, Nygaard IE, Wilken J, Brandt D, Janz KF. Postoperative activity restrictions: any evidence? Obstet Gynecol. 2006 Feb;107(2 Pt 1):305-9. doi: 10.1097/01.AOG.0000197069.57873.d6. PMID 16449116
- [Result] Winkelman WD, Erlinger AL, Haviland MJ, Hacker MR, Rosenblatt PL. Survey of Postoperative Activity Guidelines After Minimally Invasive Gynecologic and Pelvic Reconstructive Surgery. Female Pelvic Med Reconstr Surg. 2020 Dec 1;26(12):731-736. doi: 10.1097/SPV.0000000000000697. PMID 30707119
- [Result] Mueller MG, Kenton K. Activity Restrictions After Gynecologic Surgery. Obstet Gynecol. 2024 Mar 1;143(3):378-382. doi: 10.1097/AOG.0000000000005501. Epub 2024 Jan 11. PMID 38207325